CLINICAL TRIAL: NCT05120453
Title: Assessment of the Interplay Between Self-critisim and Symptom Severity Over the Course of In-patient Psychotherapeutic Treatment
Brief Title: Interplay of Self-Criticism and Symptom Severity Over the Course of In-patient Psychotherapeutic Treatment
Acronym: InSeCur
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Simone Jennissen, Principal Investigator, University Hospital Heidelberg
Other Study IDs: ST-TDEQSCL-2021
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Self-Criticism; Psychological Distress; In-Patient Treatment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the interplay between self-criticism and symptom severity in patients undergoing psychotherapeutic treatment.

DETAILED DESCRIPTION:
Participants are recruited at the University Clinic Heidelberg at the beginning of their (usually) 8-week in-patient treatment, consisting of somatic and psychotherapeutic aspects. After informed consent, patients routinely fill out weekly questionnaires about their self-criticism and their symptom severity. The overall aim of this study is to disentangle stable (between-person) effects of both self-criticism and symptom severity from within-person effects happening over time in order to better understand what drives what, or in other words, their dynamic interplay. The analysis is based on the weekly assessment of the patients. All patients receive the standard care of the in-patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing in-patient treatment at the University Clinic Heidelberg (Klinik für Allgemeine Innere Medizin und Psychosomatik)

Exclusion Criteria:

* none

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients undergoing in-patient treatment at the university clinic Heidelberg. The psychosomatic clinic treats patients over the course of (usually) 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 2778 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
SCL-K11 | Weekly Assessments over the course of the in-patient treatment (usually about 8 weeks)
  Symptom Check-List German Short Version with 11 Items
TDEQ-12 (Subscale Self-Criticism | Weekly Assessments over the course of the in-patient treatment (usually about 8 weeks)
  Theoretical Depressive Experiences Questionnaire German Short Version with 12 Items: Subscale Self-Criticism

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Dinger, Prof, Study Chair — University Hospital Heidelberg

IPD SHARING:
Plan to Share IPD: No